CLINICAL TRIAL: NCT04674540
Title: Investigation on the Cognition and Implementation of Sedation and Analgesia in EICU Critically Ill Patients
Brief Title: EICU Analgesia and Sedation Cross-sectional Survey
Acronym: EASY
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-037
Record Dates: First submitted 2020-06-15; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Sedation and Analgesia; ICU
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sedation and Analgesia Implementation Status Group: To investigate the implementation status of sedation and analgesia in ICU critical patients.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
Sedation and analgesia is a very important part of the comprehensive treatment of critically ill patients. The comprehensive management strategy of sedation and analgesia in the Intensive Care Unit (ICU) and the control of infection, the application of antibiotics, and active recovery-are equally important. Effective sedation and analgesia assessment tools and reasonable comprehensive management strategies can not only improve patient comfort, reduce discomfort memory, but also reduce nursing workload and improve clinical outcomes. The "eCASH" theory proposed by Vincent et al. in 2016 further improved the comprehensive management strategy for sedation and analgesia. Its main contents are early analgesia to make patients comfortable, minimal sedatives and maximum humanitarian care. However, unreasonable sedation, especially early deep sedation, is closely related to the poor prognosis of patients. With the update of the ICU sedation and analgesia guidelines and the continuous progress of related research, ICU doctors have gradually deepened their understanding of sedation and analgesia. At present, the level of emergency ICU development in various regions of the country is uneven, and the implementation of sedation and analgesia may also vary greatly. Therefore, by investigating and understanding the implementation of emergency ICU or ICU sedation and analgesia in various regions of the country, you can indirectly understand the familiarity of medical staff with sedation and analgesia guidelines, and formulate corresponding strategies for specific situations, which may help improve critical illness. The level of sedation and analgesia of the patient improves the treatment effect.

So far, there are few domestic research reports on the implementation of sedation and analgesia in critical patients, especially the data in the emergency ICU. This study intends to investigate the implementation status of sedation and analgesia in critically ill patients in ICU, to understand the familiarity of medical staff with sedation and analgesia guidelines, and provide a basis for further measures.

DETAILED DESCRIPTION:
Part 1: Cognitive survey

Participants: emergency and critical illness medical staff (doctors and nurses) of participating units. The number of medical staff in each unit is at least 12, among which doctors and nurses are ≥6 (the ratio is ≥3 for elementary level and ≥3 for intermediate and above).

Investigate awareness of sedation and analgesia guidelines.

Part 2: Current status of sedation and analgesia

Participants: patients older than 18 years old in the ICU of the participating unit.

1. Collect general information of patients that meet the inclusion criteria, including the patient's gender, age, body mass index (BMI), length of stay in ICU (days, with 1 effective decimal), diagnosis, acute physiology and chronicity on day 1 Health status score (Acute Physiology and Chronic Health Evaluation II, APACHE II), whether to receive mechanical ventilation, whether to use vasoconstrictor to maintain blood pressure and other information;

2. Assess whether the patients need sedation and analgesia, and divide the patients into groups.

1. Sedation assessment: Use the Richmond Sedation and Restlessness Score (RASS score) for sedation assessment. For mechanically ventilated patients, if the RASS score is ≥1, sedation is considered necessary; for patients without mechanical ventilation, if the RASS score is ≥2, consider Sedation is needed; for patients who have been given sedation and the RASS score reaches the target, sedation is also considered necessary.
2. Analgesia evaluation: The digital pain scoring method is used for awake patients, and when the score is ≥4 points, the drug is administered according to the WHO three-step analgesic principle; non-conscious patients should use the Critical-Care Pain Observation Tool (CPOT), If CPOT ≥ 3 points, it is considered that there is pain, and analgesia is needed; for patients who are already on analgesia treatment and the pain score reaches the standard, it is also considered that analgesia is needed.
3. Evaluation of delirium: Has delirium occurred after entering the ICU? Do you use delirium assessment tools? Record the means of delirium management;

3. If sedation and analgesia is required, relevant information will be collected according to the actual situation of each research unit. For patients who do not require sedation and analgesia after the second step assessment, there is no need to collect sedation and analgesia information. This information includes:

1. Is there any sedation and analgesia?
2. Information about sedation: Are sedation assessment tools used (if used, what kind of sedation assessment tools are used); are sedation target values set (record specific values)? Actual sedation score; name and dose of sedative drugs;
3. Analgesia-related information: whether to use analgesia evaluation tools (if used, what analgesia evaluation tools are recorded); whether to set an analgesia target value (record the specific value)? Actual analgesic score; name and dosage of analgesic drugs;

ELIGIBILITY:
Inclusion Criteria:

* Multiple intensive care units (ICU) and emergency intensive care units (EICU) in China
* Patients older than 18 years in the ICU/EICU

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient older than 18 years admitted to the ICU, in the participating hospitals, will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 1195 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Cognition of Sedation and Analgesia | 1 day
  Awareness of sedation and analgesia guidelines. The questionnaire involves 20 questions about the main principles and knowledge of ICU sedation and analgesia treatment.
Sedation assessment: Richmond Agitation and Sedation Scale | 1 day
  Sedation assessment: Richmond Agitation and Sedation Scale (RASS, score from -5 to 4) for sedation assessment.
Analgesia evaluation: The digital pain scoring method | 1 day
  Analgesia evaluation: The digital pain scoring method is used for awake patients (score from 0 to 10);
Analgesia evaluation: Critical-Care Pain Observation Tool | 1 day
  Analgesia evaluation: non-conscious patients should use the Critical-Care Pain Observation Tool (CPOT, score from 0 to 8).
Analgesia evaluation-Confusion Assessment Method of the Intensive Care Unit | 1 day
  Evaluation of delirium: Confusion Assessment Method of the Intensive Care Unit (CAM-ICU) for delirium evaluation.

SECONDARY OUTCOMES:
General information of patients-gender | 1 day
  gender (male or female)
General information of patients-age | 1 day
  Age (older than 18 years )
General information of patients-BMI | 1 day
  height(kg), weight(cm); weight and height will be combined to report BMI in kg/m^2).
General information of patients-length of stay in ICU | 1 day
  length of stay in ICU (day)
General information of patients-APACHE II | 1 day
  Acute Physiology and Chronic Health Evaluation II (APACHE II)

CONTACTS AND LOCATIONS:
Overall Officials: Mao Zhang, MD, Study Chair — Second Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine & Institute of Emergency Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
Need to be approved by the ethics committee

REFERENCES:
- [Background] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Background] Chanques G, Jaber S, Barbotte E, Violet S, Sebbane M, Perrigault PF, Mann C, Lefrant JY, Eledjam JJ. Impact of systematic evaluation of pain and agitation in an intensive care unit. Crit Care Med. 2006 Jun;34(6):1691-9. doi: 10.1097/01.CCM.0000218416.62457.56. PMID 16625136
- [Background] Payen JF, Bosson JL, Chanques G, Mantz J, Labarere J; DOLOREA Investigators. Pain assessment is associated with decreased duration of mechanical ventilation in the intensive care unit: a post Hoc analysis of the DOLOREA study. Anesthesiology. 2009 Dec;111(6):1308-16. doi: 10.1097/ALN.0b013e3181c0d4f0. PMID 19934877
- [Background] Jacobi J, Fraser GL, Coursin DB, Riker RR, Fontaine D, Wittbrodt ET, Chalfin DB, Masica MF, Bjerke HS, Coplin WM, Crippen DW, Fuchs BD, Kelleher RM, Marik PE, Nasraway SA Jr, Murray MJ, Peruzzi WT, Lumb PD; Task Force of the American College of Critical Care Medicine (ACCM) of the Society of Critical Care Medicine (SCCM), American Society of Health-System Pharmacists (ASHP), American College of Chest Physicians. Clinical practice guidelines for the sustained use of sedatives and analgesics in the critically ill adult. Crit Care Med. 2002 Jan;30(1):119-41. doi: 10.1097/00003246-200201000-00020. No abstract available. PMID 11902253